CLINICAL TRIAL: NCT04796623
Title: A Open-label, Multicenter Phase II Study of TQB3616 Capsules Combined With Fulvestrant Injection in Subjects With HR-positive, HER2-negative Advanced Breast Cancer
Brief Title: A Study of TQB3616 Capsules Combined With Fulvestrant Injection in Subjects With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-II-01
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: HR-positive, HER2-negative Advanced Breast Cancer
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3616 capsules combined with fulvestrant injection (Experimental): TQB3616 capsules 180 mg given orally, once daily in 28-day cycle. Fulvestrant injection was given at a fixed dose of 500mg on day 1, day 15 of the first cycle and day 1 of each subsequent cycle, and each cycle is 28 days.
  Interventions: Drug: TQB3616 capsules; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: TQB3616 capsules — TQB3616 capsules 180 mg given orally, once daily in 28-day cycle.
Drug: Fulvestrant injection — Fulvestrant injection was given at a fixed dose of 500mg on day 1, day 15 of the first cycle and day 1 of each subsequent cycle, and each cycle is 28 days.

SUMMARY:
This study is a multicenter, open-label, multi-cohort phase II clinical trials to evaluate the efficacy and safety of TQB3616 capsules combined with Fulvestrant injection in subjects with HR-positive and HER2-negative advanced and/or metastatic breast cancer, including Cohort 1 and Cohort 2. Each cohort will enroll 30-60 cases.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understood and signed an informed consent form. 2.Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months. 3. Histopathologically confirmed HR positive and HER2 negative advanced or metastatic breast cancer. 4.Cohort 1: patients had received ≤1 line of treatment. 5.Cohort 2: patients had not previously received systemic antitumor therapy. 6.Has at least one measurable lesion according to RECIST1.1 criteria. 7.Adequate laboratory indicators.

Exclusion Criteria:

* 1. Concomitant disease and medical history:

  1. Has other malignant tumors within 3 years;
  2. Has multiple factors affecting oral medication;
  3. Unalleviated toxicity ≥ grade 1 due to any previous anticancer therapy;
  4. Has active or uncontrolled severe infections before the first dose;
  5. Cirrhosis, active hepatitis#
  6. Have a history of immunodeficiency; 2. Tumor-related symptoms and treatment:

  <!-- -->

  1. Has central nervous system metastases (CNS) and/or cancerous meningitis or leptomeningeal carcinomatosis;
  2. Had received chemotherapy within 3 weeks prior to the first dose, and had received radiotherapy , hormone therapy, or other anti-tumor therapy within 2 weeks prior to the first dose;
  3. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.

     3. Has known to be allergic to Fulvestrant injection , TQB3616 or any excipient.

     4. Has Participated in other clinical trials within 4 weeks before first dose. 5. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by investigator | Baseline up to 24 months
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR), recorded from the first dose until the first documented progressive disease (PD) or death from any cause, based on investigator.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Baseline up to 24 months
  PFS defined as the time from first dose until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | Baseline up to 24 months]
  OS defined as the time from first dose to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Clinical benefit rate (CBR) | Baseline up to 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | Baseline up to 24 months
  The time when the participants first achieved complete or partial remission to disease progression.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Gansu Provincial Hostipal, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Affiliated Cancer Hospital, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang